CLINICAL TRIAL: NCT00683462
Title: An Exploratory Trial of AZD3480 (TC-1734) for the Treatment of Adult Attention-Deficit/Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Targacept Inc. (Industry)
Responsible Party: Hans-Göran Hårdemark, MD, PhD, Medical Science Director AZD3480, AstraZeneca R&D, Södertälje
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TC-1734-226-CRD-005; NCT00683215 (obsolete NCT alias)
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2009-10-30 (Estimated); Status verified 2009-10

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — ispronicline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Placebo Comparator)
  Interventions: Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: AZD3480
- 3 (Experimental)
  Interventions: Drug: AZD3480

INTERVENTIONS:
Drug: Placebo
  Arms: 1
Drug: AZD3480 — Capsules 5 mg/day (once a day) for 2 weeks
  Arms: 2
Drug: AZD3480 — Capsules 50 mg/day (once a day) for 2 weeks
  Arms: 3

SUMMARY:
A 3-way cross-over trial of two weeks of treatment with three drug conditions. AZD3480 will be given in doses of (A) 5mg/day, (B) 50 mg/day and (C) placebo to 24 non-smoking adults with DSM-IV confirmed ADHD. Three week washout between each treatment period. CYP2D6 genotyping will be completed at screening and slow metabolisers will be excluded from participation in this study. Cognitive, ADHD symptom, safety and pharmacokinetic (PK) assessments will be made during each treatment period. Safety and tolerability assessments will be a major component of the trial and all serious adverse events (SAE) will be immediately (within 24 hours) reported to both Targacept and to AstraZenca.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of DSM-IV ADHD
* Score of equal or more than 2 on at least six of nine items in at least one of the subscales of the Connor´s Adult ADHD Rating Scale (CAARS-INV)
* Score of equal or more than 4 (at least moderate severity) on the Clinical Global Impressions-Severity (CGI-S) test

Exclusion Criteria:

* Current DSM-IV Axis I psychiatric disorder (other than ADHD)
* Current user of cigarettes or other nicotine-containing product.
* Slow metabolizers as indicated by CYP2D6 genotyping.
* Use of drugs affecting cognitive function within 8 weeks prior to enrollment visit or intended use during the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-05; Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The Total Symptoms Scale Score (of ADHD) of the Connors Adult ADHD Rating Scale-Investigator Rating (CAARS-INV). | Visit 1, 2, 3, 4, 5, 8, 9, 10,13, 14 and 15

SECONDARY OUTCOMES:
Clinical Global Impressions Scales (NIMH 1985) | Visit 1, 2, 3, 4, 5, 8, 9, 10, 13, 14,15
CDR computerized cognitive battery | 2, 3, 5, 8, 10, 13, 15
CNRU computerized cognitive battery | 2, 3, 5, 8, 10, 13, 15

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Burlington, Vermont, United States

REFERENCES:
- [Derived] Potter AS, Dunbar G, Mazzulla E, Hosford D, Newhouse PA. AZD3480, a novel nicotinic receptor agonist, for the treatment of attention-deficit/hyperactivity disorder in adults. Biol Psychiatry. 2014 Feb 1;75(3):207-14. doi: 10.1016/j.biopsych.2013.06.002. Epub 2013 Jul 12. PMID 23856296